CLINICAL TRIAL: NCT03684434
Title: Development and Evaluation of a Brief Online Motivational Interviewing Intervention for Enhancing Engagement in Internet-delivered Cognitive Behaviour Therapy
Brief Title: Online Cognitive Behaviour Therapy for Depression and Anxiety: Randomized Controlled Trial Varying Treatment Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-084
Record Dates: First submitted 2018-09-11; First posted 2018-09-25 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Internet-delivered cognitive behaviour therapy; Motivational Interviewing; Randomized controlled trial; Pre-treatment; Mental health system
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online MI plus Online CBT (Experimental): An online motivational interviewing (MI) lesson will first be delivered to clients. The MI lesson is expected to take one hour to complete. No therapist support will be provided during this component of treatment. An 8-week Internet-delivered cognitive behavioural therapy (ICBT) will be then delivered to clients following completion of online MI. Clients will receive weekly support in the form of emails and phone calls from registered social workers, psychologists or supervised graduate students, who have experience delivering ICBT. Therapist will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Online MI plus Online CBT
- Online CBT (Active Comparator): An 8-week Internet-delivered cognitive behavioural therapy (ICBT) will be delivered to clients. Clients will receive weekly support in the form of emails and phone calls from registered social workers, psychologists or supervised graduate students, who have experience delivering ICBT. Therapist will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Online CBT

INTERVENTIONS:
Behavioral: Online MI plus Online CBT — An online motivational interviewing (MI) lesson will first be delivered to clients. The MI lesson is expected to take one hour to complete. No therapist support will be provided during this component of treatment. An 8-week Internet-delivered cognitive behavioural therapy (ICBT) will be then delivered to clients following completion of online MI. Clients will receive weekly support in the form of emails and phone calls from registered social workers, psychologists or supervised graduate students, who have experience delivering ICBT. Therapist will spend approximately 15 minutes per week/per client.
  Other Names: Planning for Change Lesson plus Wellbeing Course
  Arms: Online MI plus Online CBT
Behavioral: Online CBT — An 8-week Internet-delivered cognitive behavioural therapy (ICBT) will be delivered to clients. Clients will receive weekly support in the form of emails and phone calls from registered social workers, psychologists or supervised graduate students, who have experience delivering ICBT. Therapist will spend approximately 15 minutes per week/per client.
  Other Names: Wellbeing Course
  Arms: Online CBT

SUMMARY:
Anxiety and depression are prevalent and disabling conditions. Although cognitive behaviour therapy (CBT) has been shown to significantly reduce symptoms of anxiety and depression, access to the service is limited. Internet-delivered cognitive behaviour therapy (ICBT) represents a novel approach to overcoming access barriers and involves delivering therapeutic content to manage symptoms via structured online lessons. The Online Therapy Unit has been studying the efficacy of ICBT for anxiety and depression and found that ~75% of clients complete treatment and demonstrate large improvement in symptoms. However, recent research suggests that younger clients and clients with higher baseline distress are more likely to dropout of ICBT. While it remains unclear why these clients are more susceptible to attrition, it is plausible that they are experiencing a greater degree ambivalence to change and, thus, terminate treatment as a result. Motivational interviewing (MI) aims to help facilitate clients' intrinsic motivation to change by resolving ambivalence. MI has been integrated into CBT for anxiety to overcome similar concerns of poor treatment retention. Evidence suggests that the integration of MI and CBT further enhances response and completion rates. In the context of online therapy, however, the efficacy of MI remains unclear. In the current trial, the investigators aimed to assess a recently developed online MI pre-treatment (i.e., the Planning for Change lesson). A total of 480 clients (original aim for sample size was 300) applying to transdiagnostic ICBT in routine care were randomly assigned to receive the MI pre-treatment or no pre-treatment (i.e., a waiting period) prior to participating in ICBT (i.e., the Wellbeing Course). The investigators sought to examine: how ICBT with MI compared to standardized ICBT in terms of symptom change, rates of reliable improvement, intervention usage (e.g., number of lessons completed), frequency of motivational language in the first two emails to therapist, and motivation levels. It was hypothesized that there would be a small but significant effect of MI on these variables. Additionally, the investigators aimed to explore if age and severity of baseline distress moderate the effect between MI and ICBT outcomes. Younger clients and clients with higher baseline distress are more likely to drop out of ICBT and, thus, it was further hypothesized that online MI will have a greater impact on these groups.

ELIGIBILITY:
Inclusion Criteria:

* is 18 years of age or older
* is a resident of Saskatchewan, Canada
* is experiencing at least mild to moderate symptoms of anxiety and/or depression
* has not been hospitalized within the last year for mental health and/or suicide risk concerns
* is not seeking regular face-to-face therapy for anxiety and/or depression
* has access to a secure computer and the Internet
* is comfortable using technology
* is available to work through treatment each week
* is willing to provide a medical contact as emergency contact

Exclusion Criteria:

* is younger than 18 years of age
* is not a resident of Saskatchewan, Canada
* is experiencing no symptoms of anxiety and/or depression
* has been hospitalized within the last year for mental health and/or suicide risk concerns
* has unmanaged problems with alcohol, drugs, psychosis, or mania
* is seeking regular face-to-face therapy for anxiety and/or depression
* does not have access to a secure computer and the Internet
* is not comfortable using technology
* is not available to work through treatment each week
* is not willing to provide a medical contact as an emergency contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Change in motivation levels | Baseline and week 1
  Change Questionnaire - 3 Item: Items are summed into a total score. Total score ranges from 0 to 30, with higher scores representing greater self-reported levels of motivation.
Change in depression symptoms | Baseline, weeks 2, 3, 5, 6, 8, 10, 13, 25, and 53
  Patient Health Questionnaire - 9 Item: Items are summed into a total score. Total score ranges from 0 to 27, with higher scores representing more severe self-reported levels of depression.
Change in anxiety symptoms | Baseline, weeks 2, 3, 5, 6, 8, 10, 13, 25, and 53
  Generalize Anxiety Disorder - 7 Item: Items are summed into a total score. Total score ranges from 0 to 21, with higher scores representing more severe self-reported levels of anxiety.
Client engagement in online therapy (i.e., the Wellbeing Course) | week 10
  Measured by: Number of lessons completed, number of lesson logins, number of days of access, number of emails sent to therapist, number of phone calls with therapist, number of emails from therapist to client
Client feedback questions | week 1 (following completion of the Planning for Change lesson)
  Administered to only those participants assigned to the Online MI plus ICBT group: A series of rating and open-ended questions developed by the investigators designed to ascertain clients' perceptions of the Planning for Change lesson. Questions are designed to provide both quantitative and qualitative information, and do not include total scores.
Change in motivation to engage in treatment | Monday of week 1 and Sunday of week 1
  Two questions developed by Titov et al. (2010) to measure motivation to engage in ICBT: Both questions are rated on a 1 to 9 scale, with higher scores representing greater self-reported motivation levels. Questions will be independently assessed and, thus, there will be no total score.

SECONDARY OUTCOMES:
NOTE ABOUT SECONDARY MEASURES | weeks 1 to 53
  Below secondary outcome measures are routinely given in the Online Therapy Unit but were not of primary interest in the current study.
Change in panic symptoms | Weeks 2, 10, 13, 25, and 53 **Not used as a secondary measure anymore because PDSS was mistakenly not administered at baseline
  Measured by Panic Disorder Severity Scale-Self Report: Items are summed into a total score. Total scores range between 0 and 28, with higher scores representing more severe self-reported symptoms of panic.
Change in social anxiety symptoms | Weeks 2, 10, 13, 25, and 53 **Not used as a secondary measure anymore because SIAS was mistakenly not administered at baseline
  Measured by Social Interaction Anxiety Scale - 6 Item: Items are summed into a total score. Total scores range between 0 and 24, with higher scores representing more severe self-reported symptoms of social anxiety.
Change in social phobia symptoms | Weeks 2, 10, 13, 25, and 53 **Not used as a secondary measure anymore because SPS was mistakenly not administered at baseline
  Measured by the Social Phobia Scale - 6 Item: Items are summed into a total score. Total scores range between 0 and 24, with higher scores representing more severe self-reported symptoms of social phobia.
Change in quality of life symptoms | Weeks 2, 10, 13, 25, and 53 **Not used as a secondary measure anymore because EQ-5D-5L was mistakenly not administered at baseline
  Measured by EQ-5D-5L: Items are summed into six sub-total scores. The first five sub-total scores respectively assess various domains of quality of life (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each of the five sub-total scores range between 1 and 5, with higher scores representing greater self-reported severity and impairment in these various domains. The last sub-total score provides an overall index of health and can range between 0 and 100, with higher scores representing better self-reported health.
Psychological Distress | Baseline, weeks 2, 10, 13, 25, and 53 **K10 outcomes were only collected for half the sample during baseline due to the measure accidentally not being included at the start of recruitment. As such, distress was measured using the PHQ-9 and GAD-7 instead.
  Measured by the Kessler Psychological Distress Scale: Items are summed into a total score. Total scores range between 0 and 50, with higher scores representing more severe self-report psychological distress.
Change in disability | Baseline, weeks 2, 10, 13, 25, and 53
  Measure by Sheehan Disability Scale-3 Item: Items are summed into a total score. Total scores range between 0 and 30, with higher scores representing greater impairment associated with symptoms.
Change in post-traumatic symptoms | Baseline, weeks 13, 25, and 53
  Measured by Modified Brief Life Events Checklist: The Modified Brief Life Events Checklist consists of two sections. The first section assesses for exposure to a traumatic event using a checklist question. If the client endorses exposure to a traumatic event, they are provided the second section, which assesses severity of trauma symptoms. Items are summed into a total score, which can range between 0 and 80. Higher scores represent more severe self-reported symptoms of trauma.
Changes in treatment costs | Baseline, week 13, 25, and 53 **Only used to assess for group differences at baseline**
  Measured by Treatment Inventory of Costs in Psychiatric Patients (TIC-P) Adapted for Canada: A series of yes and no, rating, and frequency questions that are designed to ascertain the volume of medical consumption and productivity losses associated with mental health problems. Questions are independently analyzed and, therefore, the TIP-C does not include a total score.
Change in treatment credibility | Baseline and week 10
  Measured by Treatment Credibility Questionnaire: Items are summed into a total score. Total scores range between 3 and 27, with higher scores representing greater perceptions of ICBT credibility.
Therapeutic alliance | week 10
  Measured by Working Alliance Inventory-Short Form: Scores are summed into three sub-total scores, which respectively assess various domains of the therapeutic relationship (i.e., goal, task, and bond). Sub-total scores each range between 5 and 20, with higher scores representing better therapeutic relationship in each of the three domains assessed.
Satisfaction with Wellbeing Program assessed by the Internet-CBT Treatment Satisfaction Measure | week 10
  Measured by Internet-CBT Treatment Satisfaction Measure: A series of yes and no, rating, and open-ended questions developed by the investigators' collaborators. These questions are designed to ascertain clients' satisfaction with the Wellbeing Course and include questions, for example, that pertain to the likelihood of recommending the Wellbeing Course to a friend and whether they learned useful information throughout the course. Questions are designed to provide both quantitative and qualitative information, and do not include a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, Regina, Saskatchewan, Canada